CLINICAL TRIAL: NCT06194539
Title: The Assessment of Fertility in Men With Spinal Muscular Atrophy (SMA)
Brief Title: Assessing the Fertility Status of Men With Spinal Muscular Atrophy (SMA)
Status: Recruiting | Type: Observational
Sponsor: Bar-Chama, Natan, M.D. (Other)
Responsible Party: Sponsor
Other Study IDs: ML44640
Record Dates: First submitted 2023-11-30; First posted 2024-01-08 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2023-12

CONDITIONS: Fertility Issues
Keywords: Men; Spinal Muscular Atrophy
MeSH Terms: conditions — Infertility; Multiple Endocrine Neoplasia Type 1; Muscular Atrophy, Spinal

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will aim to assess the fertility status of men with Spinal Muscular Atrophy (SMA) not on disease-modifying therapies.

Participants will:

1. Complete online questionnaires that will assess SMA diagnosis and disease burden, medical and surgical history, medication usage, and fertility status and perspectives.
2. Over the 3-month initial study baseline period participants will provide two separate ejaculates for semen analysis and a single determination of sperm quality using DNA fragmentation testing using home collection and subsequent shipment to a central laboratory.
3. Over the initial study baseline period of 3 months study participants will obtain a blood test to determine male reproductive hormone levels.

During the 24-month study duration, participants will be requested to undergo a yearly semen analysis and complete online relevant questionnaires.

DETAILED DESCRIPTION:
Study participants will:

1. Complete online questionnaires that will assess SMA diagnosis and disease burden, medical and surgical history, medication usage, and fertility status and perspectives.
2. Over the 3-month initial study baseline period participants will provide two separate ejaculates for semen analysis and a single determination of sperm quality using DNA fragmentation testing using home collection and subsequent shipment to a central laboratory.
3. Over the initial study baseline period of 3 months study participants will obtain a blood test to determine male reproductive hormone levels.

During the 24-month study duration, participants will be requested to undergo a yearly semen analysis and complete online relevant questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form (or assent)
* Male and age greater than 18 years and less than 50 years of age with a confirmed diagnosis of SMA at the time of signing the Informed Consent Form (or assent)
* Currently not on a disease-modifying agent or therapy for SMA
* Adequately recovered from any acute illness at the time of screening, and considered clinically well enough to participate in the study.

Exclusion Criteria:

Men with a prior history of chemotherapy, radiation therapy, prostate or testicular cancer, undescended testicles and use of anabolic steroids or testosterone usage will be excluded

Ages: 18 Years to 50 Years | Sex: Male
Age Groups: Adult
Gender Based: Yes
Study Population: 75 men between the ages of 18 -50 with a diagnosis of SMA who are not on disease-modifying therapies.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Semen Volume | Two semen samples will be obtained at the initial 3 month study enrollment and then annually for the duration of the study period of 24 months
  Home collected semen ejaculates will be obtained to measure semen volume (normal > 1.5ml)
Sperm Concentration | Two semen samples will be obtained at the initial 3 month study enrollment and then annually for the duration of the study period of 24 months
  Home collected semen ejaculates will be obtained to measure sperm concentration ( normal > 15 million sperm/ml)
Sperm Motility | Two semen samples will be obtained at the initial 3 month study enrollment and then annually for the duration of the study period of 24 months
  Home collected semen ejaculates will be obtained to measure sperm motility ( normal > 39% motile sperm)
Sperm Morphology | Two semen samples will be obtained at the initial 3 month study enrollment and then annually for the duration of the study period of 24 months
  Home collected semen ejaculates will be obtained to measure sperm morphology (normal > 4% normal sperm morphology)
Sperm DNA Fragmentation Assay | At intial 3 month study enrollment
  Home collected semen ejaculates will be obtained to measure sperm DNA fragmentation rate ( normal < 30% DNA fragmented sperm)

SECONDARY OUTCOMES:
Male Reproductive Hormones - Total Testosterone Level | At intial 3 month study enrollment
  Serum total testosterone level will be obtained where normal values are 250 -1100 ng/dL
Male Reproductive Hormones - Free Testosterone Level | At intial 3 month study enrollment
  Serum free testosterone level will be obtained where normal values are 46.0 - 224.0 pg/mL
Male Reproductive Hormones - Follicle Stimulating Hormone | At intial 3 month study enrollment
  Serum FSH ( Follicle StimulatingHormone) level will be obtained where normal values are 1.6 -8.0 mIU/mL
Male Reproductive Hormones - Luteinizing Hormone | At intial 3 month study enrollment
  Serum LH ( Luteinizing Hormone) level will be obtained where normal values are 1.5- 9.3 mIU/mL
Male Reproductive Hormones - Estradiol | At intial 3 month study enrollment
  Serum Estradiol level will be obtained where normal values are < 39 pg/mL

CONTACTS AND LOCATIONS:
Overall Officials: Natan Bar-Chama, MD, Principal Investigator — The Mount Sinai Hospital
Locations (1):
- Natan Bar-Chama MD, Cresskill, New Jersey, United States